CLINICAL TRIAL: NCT04139499
Title: Use of High-resolution Manometry to Detect Upper Airway Obstruction During Sleep
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0184; SMPH/SURGERY/OTOLARYNGOLOGY (Other: UW, Madison); A539770 (Other: UW, Madison); UWF-SMPH -Funding (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; Continuous positive airway pressure (CPAP); Sleep manometry
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adults with OSA: Adults with obstruction at any or all of the four levels of interest (velopharynx, oropharynx, tongue base, epiglottis) will represent the experimental group.
  Interventions: Procedure: Drug-induced sleep endoscopy (DISE); Procedure: High-resolution manometry (HRM):
- Children with OSA: Children with obstruction at any or all of the four levels of interest (velopharynx, oropharynx, tongue base, epiglottis) will represent the experimental group.
  Interventions: Procedure: Drug-induced sleep endoscopy (DISE); Procedure: High-resolution manometry (HRM):
- Adult control: Adult without any obstruction at four levels of interest (velopharynx, oropharynx, tongue base, epiglottis) will represent a control.
  Interventions: Procedure: Drug-induced sleep endoscopy (DISE); Procedure: High-resolution manometry (HRM):
- Children control: Children exam will be done for all the participants. Subject without obstruction represent a control.
  Interventions: Procedure: Drug-induced sleep endoscopy (DISE); Procedure: High-resolution manometry (HRM):

INTERVENTIONS:
Procedure: Drug-induced sleep endoscopy (DISE) — DISE involves administering anesthetic to a patient to simulate a sleep state, and then visualizing the upper airway using transnasal flexible endoscopy. Sites of obstruction at key locations including the adenoids, soft palate, lateral oropharynx, tongue base, and epiglottis can be identified.
Procedure: High-resolution manometry (HRM): — After the necessary clinical information has been obtained (if obstruction is occurring at those levels and, if so, to what degree), a flexible high-resolution manometry (HRM) catheter will be passes through the contralateral nostril to record pressure along the length of the pharynx at those same sites.

SUMMARY:
Obstructive sleep apnea (OSA) is a major public health issue in both children and adults, present in 1-5% of children and 10-30% of adults. It is characterized by repeated episodes of airway obstruction during sleep, leading to brain arousal, sympathetic activation, oxygen desaturation, sleep fragmentation, and non-restorative sleep. Patients report daytime tiredness, insomnia, and morning headaches. Children with OSA experience daytime somnolence, difficulties at school, behavioral problems, enuresis, and reduced quality of life. If left untreated, OSA can lead to numerous complications including hypertension, cardiovascular disease, stroke, and insulin resistance. Sleep partners are also affected, with patients viewing their disorder as a burden and sleeping in separate rooms. Further, disease prevalence is increasing as obesity increases.

Continuous positive airway pressure (CPAP) is the current gold standard treatment for OSA. If used effectively and consistently, it can improve patient symptoms. However, adherence is generally poor, with patients experiencing physical discomfort, chest discomfort, and dry mouth. For those patients that cannot tolerate CPAP, surgical intervention is an option. In children, this typically starts with adenotonsillectomy. However, 20-75% of children will have persistent symptoms after adenotonsillectomy. In adults, anatomic factors including tonsil hypertrophy and redundant pharyngeal tissue can contribute to upper airway obstruction and may also necessitate higher pressures for effective CPAP treatment. Even if surgical intervention does not cure the OSA, it may make CPAP more tolerable and improve CPAP adherence.

Sleep-related airway obstruction is a complex phenomenon potentially involving multiple anatomic levels. For patients with persistent symptoms despite initial therapy or intolerance to CPAP, further evaluation of the upper airway is clinically valuable. Polysomnography (PSG) is the gold standard for diagnosing OSA, but it does not provide information on the location(s) of upper airway obstruction. Knowledge of the precise sites of obstruction is critical to planning effective sleep surgery. Currently, this is accomplished with drug-induced sleep endoscopy (DISE). DISE was originally proposed in 1991 and involves administering anesthetic to a patient to simulate a sleep state, and then visualizing the upper airway using transnasal flexible endoscopy. Sites of obstruction at key locations including the adenoids, soft palate, lateral oropharynx, tongue base, and epiglottis can be identified.

Though DISE offers valuable clinical information, it has notable limitations. First, it cannot evaluate the entire upper airway simultaneously, as any obstruction occurring superiorly precludes visualization of any obstruction occurring more inferiorly. Second, interpretation of DISE is subjective and there is no universally accepted system for analysis. Rating systems are qualitative, using grades such as complete, partial, or no obstruction as opposed to quantitative measurements.

The optimal sleep assessment would be quantitative, reliable, and provide information on the entire upper airway simultaneously. A potential alternative to DISE which could meet these criteria is sleep manometry. Measurement of upper airway pressures captures the effects of obstruction along the entire upper airway, from the nasopharynx to larynx. Prior studies have attempted to employ manometry, but have been limited primarily by inadequate equipment and suboptimal methods of data analysis. Woodson et al. used a solid-state manometer with diameter of 2.3 mm and 5 sensors to detect palatal obstruction and tongue base obstruction in patients with OSA. They also used the same approach to detect persistent tongue base obstruction following uvulopalatopharyngoplasty. While these studies help demonstrate that manometry can be a useful adjunct to OSA assessment, they are severely limited both by the type of manometer used as well as the lack of a clear, detailed description of the method of data analysis.

High-resolution manometry (HRM) uses pressure censors spaced 1 cm apart to allow for pressure measurement along the entire upper airway. The investigators have previously applied HRM to assessment of swallow physiology. Sophisticated methods of automated data analysis have been developed that have been shown to be reliable for both expert and novice users . Further, pattern recognition techniques have been applied to identify dysphagia and specific swallowing abnormalities. Application of this technology and modification of existing data analysis platforms will allow for a quantitative, reliable, and comprehensive assessment of upper airway obstruction during sleep in both children and adults, with potential for development of algorithms to predict effects of targeted surgical therapy at all levels of the upper airway.

ELIGIBILITY:
Inclusion Criteria:

ADULTS

* Age 18-90
* Any participant undergoing sleep endoscopy as part of standard clinical care would be eligible. This entails physician concern for sleep-disordered breathing and corresponding questionnaire and/or polysomnogram results supporting a diagnosis of obstructive sleep apnea.
* Participants without apnea are eligible, provided they are undergoing tonsillectomy or bronchoscopy for either chronic tonsillitis or airway assessment without concern for history of sleep apnea.
* Women with childbearing potential will not be excluded, as the proposed experiment would have no potential ramifications on childbearing potential.

CHILDREN

* Age 5-17
* Any patients undergoing sleep endoscopy as part of standard clinical care would be eligible.
* Participants undergoing either tonsillectomy for chronic tonsillitis or bronchoscopy for airway assessment.
* Women with childbearing potential will not be excluded, as the proposed experiment would have no potential ramifications on childbearing potential.

Exclusion Criteria:

* Participant desire to avoid added anesthesia time.
* Inability to safely tolerate the added anesthesia time (about 5-10 minutes) for the experiment (as judged by either otolaryngologist or anesthesiologist).
* Pregnant women
* Vulnerable groups (i.e., prisoners, individuals lacking consent capacity, individuals unable to read the consent form).

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Majority of subjects will be those children and adults who will be undergoing DISE as part of their standard clinical care.
  However, it is desirable to have cleaner controls without obstruction at any level to confirm that the visual absence of obstruction also represents a manometrically normal respiration. Thus, subjects without symptoms of obstructive sleep apnea who are undergoing a surgical procedure will be recruited. Simultaneous performance of DISE (to confirm no obstruction) and HRM in such subjects would take about 5 minutes. Further, the time required is within the variability typically expected at an academic center where trainees may participate in cases.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Baseline pressure at different levels of obstruction in OSA participants as measured by HRM | Up to 24 hour
  Baseline pressure at different levels of obstruction in OSA participants will be measured by HRM. The aim is to determine if HRM can identify obstruction at the velopharynx, oropharynx, tongue base, and epiglottis as seen on DISE. obstruction at each site will be identified on DISE. Subject data will be divided into three groups for each site based on results from the DISE exam, which are currently used clinically: no obstruction (<50% obstructed), partial obstruction (50-75% obstruction), or complete obstruction (>75% obstruction). Investigator will be checking if values differ across the three categories of obstruction.
Maximum pressure at different levels of obstruction in OSA participants as measured by HRM | Up to 24 hour
  Maximum pressure at different levels of obstruction in OSA participants will be measured by HRM. The aim is to determine if HRM can identify obstruction at the velopharynx, oropharynx, tongue base, and epiglottis as seen on DISE. obstruction at each site will be identified on DISE. Subject data will be divided into three groups for each site based on results from the DISE exam, which are currently used clinically: no obstruction (<50% obstructed), partial obstruction (50-75% obstruction), or complete obstruction (>75% obstruction). Investigator will be checking if values differ across the three categories of obstruction.
Duration of pressure elevation at different levels of obstruction in OSA participants as measured by HRM | Up to 24 hour
  Duration of pressure at different regions of obstruction in OSA participants will be measured by HRM. The aim is to determine if HRM can identify obstruction at the velopharynx, oropharynx, tongue base, and epiglottis as seen on DISE. obstruction at each site will be identified on DISE. Subject data will be divided into three groups for each site based on results from the DISE exam, which are currently used clinically: no obstruction (<50% obstructed), partial obstruction (50-75% obstruction), or complete obstruction (>75% obstruction). Investigator will be checking if values differ across the three categories of obstruction.
Pressure integral at different levels of obstruction in OSA participants as measured by HRM | Up to 24 hour
  Pressure integral at different regions of obstruction in OSA participants will be measured by HRM. The aim is to determine if HRM can identify obstruction at the velopharynx, oropharynx, tongue base, and epiglottis as seen on DISE. obstruction at each site will be identified on DISE. Subject data will be divided into three groups for each site based on results from the DISE exam, which are currently used clinically: no obstruction (<50% obstructed), partial obstruction (50-75% obstruction), or complete obstruction (>75% obstruction). Investigator will be checking if values differ across the three categories of obstruction.
Number of participants identified with upper airway obstruction during sleep using DISE vs HRM | Up to 24 hour
  Number of participants identified with upper airway obstruction during sleep will be a parameter to compare the efficacy of HRM and to evaluate if HRM can compliment DISE for diagnosing the level of obstruction. Obstruction can be at the velopharynx, oropharynx, tongue base, and epiglottis
Apnea-hypopnea index (AHI) as obtained from polysomnography | Up to 24 hour
  To determine the relationship between manometric variables and standard assessment used to evaluate OSA, apnea-hypopnea index (AHI) will be obtained from polysomnography.
  AHI is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation. Combining AHI and oxygen desaturation gives an overall sleep apnea severity score that evaluates both the number of sleep disruptions and the degree of oxygen desaturation (low oxygen level in the blood).
  The AHI values for adults are categorized as:
  Normal: AHI<5 Mild sleep apnea: 5≤AHI<15 Moderate sleep apnea: 15≤AHI<30 Severe sleep apnea: AHI≥30 For children, because of their different physiology, an AHI in excess of 1 is considered abnormal. Pediatric patients presenting with AHI of 2 or greater will often be referred for treatment.
Pediatric Sleep Questionnaire score as an indicator of OSA severity | Up to 24 hour
  To determine the relationship between manometric variables and standard assessment used to evaluate OSA, Pediatric Sleep Questionnaire score will be obtained.
  This scale contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric OSA features. If eight or more statements are answered "yes", child is referred for sleep evaluation. Higher score correlates to more severe OSA.
Epworth Sleepiness Scale score as an indicator of OSA severity | Up to 24 hour
  To determine the relationship between manometric variables and standard assessment used to evaluate OSA, Epworth Sleepiness Scale score will be obtained.
  The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which participants rate their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. When they finish the test, the values are added up. The total score is based on a scale of 0 to 24. The scale estimates whether the participants are experiencing excessive sleepiness that possibly requires medical attention. Scores range from 0 to 24, having scores above 9 implicate that the person is considerably sleepy to seek medical attention.
To determine the relationship between manometric variables and STOP-BANG Sleep Apnea Questionnaire score | Up to 24 hour
  To determine the relationship between manometric variables and standard assessment used to evaluate OSA, STOP-BANG Sleep Apnea Questionnaire score will be obtained.
  The snoring, tiredness, observed apnea, high BP (STOP) and snoring, tiredness, observed apnea, high BP-BMI, age, neck circumference and gender (STOP-Bang) questionnaire consists of 8 yes/no questions.
  For general population Low risk of OSA: Yes to 0-2 questions Intermediate risk of OSA: Yes to 3-4 questions High risk of OSA: Yes to 5-8 questions or Yes to 2 or more of 4 STOP questions + male gender or Yes to 2 or more of 4 STOP questions + BMI > 35 kg/m2 or Yes to 2 or more of 4 STOP questions + neck circumference (17"/43cm in male, 16"/41cm in female)
Efficacy of manometric variables to predict which subjects benefit from surgical interventions for OSA | 2 years
  to determine if manometric variables can predict which subjects benefit from surgical interventions (performed as part of standard clinical care) based on changes in postoperative obstructive sleep apnea assessments.
Correlation between the outcome of surgery and manometric variables as assessed by the number of participants with improved Apnea-hypopnea index (AHI) after surgery | 2 years
  In this study, "improvement" in OSA symptoms will be defined as at least a 50% change in AHI or questionnaire score. Logistic regression analyses will be performed to determine if there is a difference in the aforementioned manometric parameters between patients who improve and do not improve for interventions at a given level (velopharynx, oropharynx, tongue base, epiglottis).

OTHER OUTCOMES:
Pharyngeal pressures from spontaneous saliva swallows occurring during the DISE exam in pediatric and adult subjects. | 2 years
  Data will only be analyzed from spontaneous swallows that occur while the subjects are under an anesthesia-induced sleep state. Thus, all spontaneous swallows will only be saliva swallows (i.e., no food or liquid will be delivered to the subjects, as they will be under anesthesia and any bolus swallows would not be safe).
  Manometric data will be collected during spontaneous swallows (both adults and children) and pressure variables normally calculated for awake adult swallowing will be extracted from the velopharynx, tongue base, hypopharynx, and upper esophageal sphincter regions. Data for this aim will only be analyzed descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Mcculloch, MD, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No